CLINICAL TRIAL: NCT05893108
Title: The Effect of Ethosomal Gel Bearing Losartan 5% on The Patient and Observer Scar Assessment Scale Score, Degree of Erythema and Pigmentation, Surface Area, Thickness and Pliability of Human Keloids
Brief Title: Ethosomal Gel Bearing Losartan 5% for Keloid Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuni Eka Anggraini (Other)
Collaborators: Gadjah Mada University (Other)
Responsible Party: Sponsor-Investigator, Yuni Eka Anggraini, Candidate of Doctor, Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT0012023
Record Dates: First submitted 2023-05-24; First posted 2023-06-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Keloid
Keywords: Angiotensin II; Angiotensin II blocker; 5 % Losartan Gel; 10 mg/ml Triamcinolone acetonide; Keloid
MeSH Terms: conditions — Keloid | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Two groups received different treatment at the same time. Both outcomes were measured at the same time before and after treatment with 4 measurements.
Who Masked: Outcomes Assessor
Masking Description: The treatment given to participants is not known by any of the outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan (Experimental): ethosomal gel bearing losartan 5% applied two times a day for three consecutive months on keloids
  Interventions: Drug: Ethosomal gel bearing losartan 5%
- Triamcinolone (Active Comparator): Intralesional injection of triamcinolone acetonide 10 mg/ml every two weeks for three consecutive months on keloid
  Interventions: Drug: triamcinolone acetonide 10 mg/ml

INTERVENTIONS:
Drug: Ethosomal gel bearing losartan 5% — A pharmaceutical company with a good manufacturing practice certificate is developing ethosomal gel bearing losartan 5%
  Arms: Losartan
Drug: triamcinolone acetonide 10 mg/ml — intralesional injection
  Other Names: TA 10 mg/ml
  Arms: Triamcinolone

SUMMARY:
The objectives are to compare the efficacy of pre and post-treatment and between 5% losartan potassium loaded in ethosomal gel and 10 mg/ml triamcinolone acetonide injection based on the indicator score of The patient and observer scar assessment scale 3.0 (POSAS 3.0), degree of erythema and pigmentation, area size, thickness and density of human keloids.

DETAILED DESCRIPTION:
After being informed about the study and the associated risks and benefits, participants will be randomly allocated to one of two groups, each consisting of 23 individuals. After being informed about the study and the associated risks and benefits, participants will be randomly allocated to one of two groups, each consisting of 23 individuals. One group will receive the topical application of 5% losartan gel, while the other will receive an injection of triamcinolone acetonide 10mg/ml. After being informed about the study and the associated risks and benefits, participants will be randomly allocated to one of two groups, each consisting of 23 individuals. To measure the subjective and objective changes that occur in the keloid before and after treatment, outcome assessors will be blinded. Measurements will be taken four times over the course of three months.

ELIGIBILITY:
Inclusion Criteria:

* keloid patients who came to the outpatient clinic of general hospital Syafira Pekanbaru during 2023-2024,
* age is greater than or equal to 18 year
* keloid scar than or equal to 25 cm2
* duration of keloids longer than or equal to 6 months
* no drug interventions or not currently on keloid medications for the last two months.

Exclusion Criteria:

* subjects who do not understand the rubric of The patient and observer scar assessment scale (POSAS) and were not willing to participate
* subjects with nodular keloids
* subjects within antihypertensive therapy, pregnancy, malignancy, history of allergies, active skin lesions or bleeding in the keloid area.
* subjects in the treatment of keloid within the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
The patient and observer scar assessment scale score (POSAS 3.0) | change from baseline the POSAS score at 4,8, and 12 weeks, consecutively.
  The Patient and Observer Scar Assessment Scale 3.0 consists of sixteen items of the patient questionnaire (PSAS) with maximum and minimum values are 80 and 16, consecutively; and seven items of the observer questionnaire (OSAS) with maximum and minimum values are 35 and 7, consecutively. The lower score, the better result of the keloid.

SECONDARY OUTCOMES:
Degree of erythema and hyperpigmentation | change from baseline the degree of erythema and hyperpigmentation at 4, 8 and 12 weeks, consecutively.
  The colors are taken using dermoscopy and quantifiably analysed using image analysis ImageJ
the width of the keloid surface area (mm2) | change from baseline width of keloid surface area at 4, 8 and 12 weeks, consecutively.
  The surface area is taken by digital photography and quantifiably analysed using image analysis ImageJ
The thickness of keloid (mm) | change from baseline thickness of keloid at 4, 8 and 12 weeks, consecutively.
  The thickness of the keloids is assessed using high-frequency ultrasonography
The degree of pliability of keloid (durometer unit) | change from baseline pliability at 4, 8 and 12 weeks, consecutively.
  The pliability of keloids is assessed using durometer shore type oo (Teclock Japan)

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Syafira, Pekanbaru, Riau, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in keloid treatment. Data or samples shared will be coded, with no protected health information included. Approval of the request of the dataset is prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Two years after publishing the result, the data will be provided and be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research.

REFERENCES:
- [Background] Bock O, Schmid-Ott G, Malewski P, Mrowietz U. Quality of life of patients with keloid and hypertrophic scarring. Arch Dermatol Res. 2006 Apr;297(10):433-8. doi: 10.1007/s00403-006-0651-7. Epub 2006 Mar 10. PMID 16528552
- [Background] Elsaie ML. Update on management of keloid and hypertrophic scars: A systemic review. J Cosmet Dermatol. 2021 Sep;20(9):2729-2738. doi: 10.1111/jocd.14310. Epub 2021 Jul 3. PMID 34169622
- [Background] Steckelings UM, Czarnetzki BM. The renin-angiotensin-system in the skin. Evidence for its presence and possible functional implications. Exp Dermatol. 1995 Dec;4(6):329-34. doi: 10.1111/j.1600-0625.1995.tb00056.x. PMID 8608339
- [Background] Silva IMS, Assersen KB, Willadsen NN, Jepsen J, Artuc M, Steckelings UM. The role of the renin-angiotensin system in skin physiology and pathophysiology. Exp Dermatol. 2020 Sep;29(9):891-901. doi: 10.1111/exd.14159. PMID 32697884
- [Background] Hedayatyanfard K, Ziai SA, Niazi F, Habibi I, Habibi B, Moravvej H. Losartan ointment relieves hypertrophic scars and keloid: A pilot study. Wound Repair Regen. 2018 Jul;26(4):340-343. doi: 10.1111/wrr.12648. Epub 2018 Oct 25. PMID 30099811
- [Background] Khodaei B, Nasimi M, Nassireslami E, Seyedpour S, Rahmati J, Haddady Abianeh S, Motavalli Khiavi F. Efficacy of Topical Losartan in Management of Mammoplasty and Abdominoplasty Scars: A Randomized, Double-Blind Clinical Trial. Aesthetic Plast Surg. 2022 Oct;46(5):2580-2587. doi: 10.1007/s00266-022-02935-2. Epub 2022 May 25. PMID 35614156
- [Derived] Anggraini YE, Trisnowati N, Martien R, Danarti R. A randomised clinical trial study assessing the efficacy of 5% losartan potassium loaded in ethosomal gel to treat human keloids: a trial protocol. Trials. 2024 Jan 2;25(1):12. doi: 10.1186/s13063-023-07880-2. PMID 38167064